CLINICAL TRIAL: NCT06338826
Title: Interventional, Multicenter, Open-label, Randomized, Non-comparative Trial Evaluating the Safety, in Terms of HBV Virological Control At 96 Weeks, of 2 Antiviral Treatment Relief Strategies, in Patients Co-infected with the HIV-1 and HBV Viruses
Brief Title: Study Evaluating the Safety, in Terms of HBV Virological Control At 96 Weeks, of 2 Antiviral Treatment Relief Strategies, in Patients Co-infected with the HIV-1 and HBV Viruses
Acronym: BI-LIGHT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ANRS0250s-BI-LIGHT
Record Dates: First submitted 2023-11-27; First posted 2024-04-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections; HBV Coinfection
MeSH Terms: conditions — HIV Infections | interventions — Racivir; dolutegravir

STUDY DESIGN:
Intervention Model Description: Interventional, sequential, Phase IIA equivalent, multicenter, open-label, randomized, non-comparative study evaluating, for 96 weeks, the safety in terms of HBV virological control of 2 antiviral therapy relief strategies, in HIV-1 and HBV co-infected patients with prolonged virological success (undetectable HIV-1 and HBV viral loads for ≥ 2 years) and on unmodified antiviral therapy for ≥ 1 year.
  Participants will be randomized 1:2:2 into 3 parallel arms:
  * Arm 1 (reference arm): Continuation of continuous (7 days/week) triple antiviral therapy including TDF or TAF
  * Arm 2 (T4): Relief from previous triple antiviral therapy (containing TDF or TAF) on 4 out of 7 consecutive days
  * Arm 3 (B7): Switch from prior triple antiviral therapy (containing TDF or TAF) to continuous dual therapy without TDF or TAF but including 3TC in combination with Dolutegravir (DTG) or ritonavir-boosted Darunavir (rDVR). The choice of dual therapy is left to the discretion of the investigator.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (No Intervention): - Arm 1 (reference arm): Continuation of continuous (7 days/week) triple antiviral therapy including TDF or TAF
- Arm 2 (T4): (Experimental): - Arm 2 (T4): Relief from previous triple antiviral therapy (containing TDF or TAF) on 4 out of 7 consecutive days
  Interventions: Drug: TDF - 245mg or TAF -25mg associated to 3TC - 300mg or FTC - 200mg and a NNRTI or PI/r or INSTI
- Arm 3 (B7) (Experimental): Switch from prior triple antiviral therapy (containing TDF or TAF) to continuous dual therapy without TDF or TAF but including 3TC in combination with Dolutegravir (DTG) or ritonavir-boosted Darunavir (rDVR
  Interventions: Drug: Dual therapy with 3TC in combination with DTG or ritonavir-boosted Darunavir (rDVR)

INTERVENTIONS:
Drug: TDF - 245mg or TAF -25mg associated to 3TC - 300mg or FTC - 200mg and a NNRTI or PI/r or INSTI — The study will include patients under current daily antiretroviral tritherapy not modified for ≥ 12 months must including tenofovir disoproxil fumarate (TDF) 245mg or tenofovir alafenamide fumarate (TAF -25mg) associated to lamivudine (3TC - 300mg) or emtricitabine (FTC - 200mg) and a NNRTI or PI/r or INSTI to choose from
  * NNRTI = efavirenz, rilpivirine, etravirine, doravirine
  * PI/r = atazanavir/r ou darunavir/r
  * INSTI = bictegravir, dolutegravir, elvitegravir/cobicistat, raltegravir
  Arms: Arm 2 (T4):
Drug: Dual therapy with 3TC in combination with DTG or ritonavir-boosted Darunavir (rDVR) — dual therapy without TDF or TAF but including 3TC in combination with Dolutegravir (DTG) or ritonavir-boosted Darunavir (rDVR
  Arms: Arm 3 (B7)

SUMMARY:
The main objective of this study is to evaluate at 96 weeks the safety with respect to hepatitis B control of 2 treatment reduction strategies for patients with previously controlled HIV-HBV co-infection on continuous triple therapy

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1-HBV co-infection (positive HIV-1 serology associated with 2 positive HBsAg serologies within more than 6 months);
2. Age ≥ 18 years
3. Fibroscan less than 6 months < 9kPa
4. Current daily antiretroviral tritherapy not modified for ≥ 12 months must including tenofovir disoproxil fumarate (TDF) 245mg or tenofovir alafenamide fumarate (TAF -25mg) associated to lamivudine (3TC - 300mg) or emtricitabine (FTC - 200mg) and a NNRTI or PI/r or INSTI to choose from

   * NNRTI = efavirenz, rilpivirine, etravirine, doravirine
   * PI/r = atazanavir/r ou darunavir/r
   * INSTI = bictegravir, dolutegravir, elvitegravir/cobicistat, raltegravir;
5. Absence of documented HBV and HIV genotypic resistance compromising virologic control of any of the maintenance strategies. Patients with no genotypic history may be included);
6. HIV CV < 50cp/ml for ≥ 2 years (only 1 annual blip allowed if HIV CV < 200cp/ml and previous and subsequent viral loads are undetectable);
7. HBV CV < 10 IU/ml for ≥ 2 years (only 1 annual blip allowed if HBV CV < 200IU/ml and if previous and subsequent viral loads are undetectable);
8. Have ≥ 3 available measurements of HIV CV < 50cp/ml and HBV CV < 10 IU/mL over the past 24 months (including that of pre-inclusion);
9. CD4 lymphocytes > 250/mm3 at pre-inclusion;
10. ALT < 3N at pre-inclusion;
11. For women of childbearing potential, negative pregnancy test and commitment to use effective contraception throughout the trial;
12. Person affiliated with or benefiting from a social security system;
13. Free, informed, written consent, signed by the person and the investigator at the latest on the day of inclusion and before any examination carried out as part of the study (article L1122-1-1 of the Public Health Code)

Exclusion Criteria:

1. HIV-2 infection;
2. HIV and/or HBV genotype not compatible with dual therapy DTG-3TC or DRVr-3TC;
3. HBeAg+;
4. Fibrosis history at stage F3-F4 in pre-therapy evaluated by PBH, fibrotest and/or fibroscan with a value of Elastometry ≥ 9kPa;
5. Chronic active viral hepatitis C (HCV RNA positive);
6. Delta co-infection;
7. Alcohol consumption > 14 units/week for women and 21 units/week for men;
8. Current treatment with chemo- or immunotherapy (including interferon or interleukins);
9. Active opportunistic infection or acute treatment for opportunistic infection;
10. Any condition (drug use, neurological, neuropsychiatric, etc.) that, in the judgment of the investigator, may compromise patient compliance and adherence to the protocol;
11. Pregnant or breastfeeding woman or refusal of contraception;
12. Major incapacity, legal protection, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with HBV virological failure at 96 weeks. | 96 weeks
  HBV virologoical failure is defined by 2 successive varial load ≥ 10UI/ml

SECONDARY OUTCOMES:
• HBV virological success rate at 48 weeks | at Week 48
  HBV virological success is defined by a viral load ≤10 UI/ml
• HIV virological success rate at 48 and 96 weeks | At week 48 and week 96
  HIV virological success is defined by a viral load ≤ 50 cp/ml
• Time to virological failure (rebound HBV and/or HIV viral load) | between Week 0 and Week96
• The rate of participants with at least one HBV viral load blip until W48 and until W96 | At week 48 and week 96
  a blip is defined by a HBV viral load >10UI/mL followed by a control value ≤ 10UIml
• Selection of HBV resistance mutations at the time of virological failure | between Week 0 and Week 96
• Incidence of grade 3 or higher adverse events of grade 3 or higher, incidence of adverse events and incidence of strategy discontinuation of the strategy at W48 and W96 | At week 48 and week 96
• Evolution of CD4 from W0 to W48 and W96 | Week 0 to Week 48 and week 96
• Evolution of total cholesterol from W0 to W48 and W96 | from Week 0 to Week 48 and Week 96
• Evaluation of the adherence by self-reported questionnaire | at Week 0, Week 12, Week 24, Week 48, Week 72 and Week 96
  without analysis scale
• Evaluation of quality of life using the Pro-Qol self-questionnaire | at Week 0, Week 12, Week 24, Week 48, Week 72 and Week 96
  without analysis scale
Evolution of CD8 T lymphocytes from W0 to W48 and W96 | Week 0 to Week 48 and week 96
Evolution of the CD4/CD8 ratio from W0 to W48 and W96 | Week 0 to Week 48 and week 96
Evolution of LDL-c from W0 to W48 and W96 | from Week 0 to Week 48 and Week 96
Evolution of HDL-c from W0 to W48 and W96 | from Week 0 to Week 48 and Week 96
Evolution of triglycerides from W0 to W48 and W96 | from Week 0 to Week 48 and Week 96
Evolution of fasting blood sugar from W0 to W48 and W96 | from Week 0 to Week 48 and Week 96
HBV virological success rate at 96 weeks between arms | at Week 96
  HBV virological success is defined by a viral load ≤10 UI/ml

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bottero, Principal Investigator — Bicetre Hospital

IPD SHARING:
Plan to Share IPD: Undecided